CLINICAL TRIAL: NCT00587301
Title: A Prospective, Open-label Study to Evaluate the Safety and Efficacy of Lap-Band® Adjustable Gastric Band (LAGB®) Operations in the Treatment of Morbidly Obese Adolescents (Ages 14-17)
Brief Title: Lap-Band Surgery on Adolescents for Safety and Efficacy
Acronym: ALAGB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Hope Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11876; G050010 (Other: H 11876)
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Obesity; DM
Keywords: Child Obesity
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lap-Band (Experimental): Lap-band surgery in treatment of morbidly obese adolescents
  Interventions: Device: Lap-Band

INTERVENTIONS:
Device: Lap-Band — Obesity and adolescents
  Other Names: Lap-Band Adjustable Gastric Band (LAGB) Operation

SUMMARY:
This study is to demonstrate the safety and efficacy of the use of the LAP-BAND surgery in the morbidly obese adolescent population.

DETAILED DESCRIPTION:
STUDY OBJECTIVES: Is to demonstrate the safety and efficacy of the use of the LAP-BAND® System in the morbidly obese adolescent population in the United States, and therefore provide these individuals with a significantly less morbid and reversible surgical option for weight loss.

STUDY VARIABLES:The primary efficacy variable is weight loss evaluated in terms of % excess weight loss (EWL).

DESIGN:Prospective, open-label, and single center

ELIGIBILITY:
Inclusion Criteria:

* Be at least 14 and less than 18 years of age at the time of enrollment into the study.
* Have a BMI of at least 40
* Have a history of obesity for at least 5 years, including failed attempts at diet and medical management of obesity.
* Confirmation by a psychologist or psychiatrist experienced with adolescents that the subject is sufficiently mature emotionally to comply with the study protocol.

Express willingness to follow protocol requirements.

•Assure investigators that subject, if female of childbearing potential, is using an appropriate form of contraception.

Exclusion Criteria:

* Intention or need to have another surgical procedure for weight reduction within 12 months of Lap Band placement.
* History of congenital or acquired anomalies of the G.I. tract, such as; congenital or acquired intestinal telangiectasia, Crohn's disease or ulcerative colitis; severe cardiopulmonary disease or severe coagulopathy; hepatic insufficiency or cirrhosis.
* Presence of dysphagia or documented esophageal dysmotility.
* Patients with autoimmune connective tissue disorders
* Patients with acute abdominal infections
* Pregnancy or intention of becoming pregnant in the next 12 months.
* Presence of psychiatric problems or immaturity which would compromise cooperation with the study protocol.
* History of previous bariatric surgery, intestinal obstruction or adhesive peritonitis.
* Presence of localized or systemic infection at the time of surgery.
* Chronic use of aspirin and/or non-steroidal anti-inflammatory medications and unwillingness to discontinue the use of these concomitant medications.
* History of gastric or esophageal surgery.
* Use of weigh loss medications simultaneously

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2005-06; Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Ren-Fielding, M.D., Principal Investigator — NYUSOM
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- See also: NYU Program for Surgical Weight Loss — http://nyuweightloss.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lap-Band
Started | 119
Completed | 74
Not Completed | 45
Not completed — Screen Failure | 9
Not completed — Lost to Follow-up | 22
Not completed — Withdrawal by Subject | 7
Not completed — Protocol Violation | 7

BASELINE CHARACTERISTICS:
Arm/Group | Lap-Band
Number analyzed (Participants) | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.1 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 108
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 90
  More than one race | 0
  Unknown or Not Reported | 15
Region of Enrollment [Number; unit: participants]
  United States | 119

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Excess Weight Loss (EWL)
Time Frame: Year 1
Measure: Mean (Standard Deviation); unit: percentage of EWL
Arm/Group | Lap-Band
Number analyzed (Participants) | 106
percentage of EWL | 40.88 (25.12)

2. Secondary Outcome: Body Mass Index (BMI)
Time Frame: Year 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Lap-Band
Number analyzed (Participants) | 106
kg/m^2 | 37.67 (8.93)

3. Primary Outcome: Percentage of Excess Weight Loss (EWL)
Time Frame: Year 2
Measure: Mean (Standard Deviation); unit: percentage of EWL
Arm/Group | Lap-Band
Number analyzed (Participants) | 95
percentage of EWL | 44.18 (26.36)

4. Primary Outcome: Percentage of Excess Weight Loss (EWL)
Time Frame: Year 3
Measure: Mean (Standard Deviation); unit: percentage of EWL
Arm/Group | Lap-Band
Number analyzed (Participants) | 87
percentage of EWL | 45.19 (25.13)

5. Primary Outcome: Percentage of Excess Weight Loss (EWL)
Time Frame: Year 4
Measure: Mean (Standard Deviation); unit: percentage of EWL
Arm/Group | Lap-Band
Number analyzed (Participants) | 81
percentage of EWL | 42.96 (26.30)

6. Primary Outcome: Percentage of Excess Weight Loss (EWL)
Time Frame: Year 5
Measure: Mean (Standard Deviation); unit: percentage of EWL
Arm/Group | Lap-Band
Number analyzed (Participants) | 74
percentage of EWL | 42.6 (26.66)

7. Secondary Outcome: Body Mass Index (BMI)
Time Frame: Year 2
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Lap-Band
Number analyzed (Participants) | 95
kg/m^2 | 36.54 (9.10)

8. Secondary Outcome: Body Mass Index (BMI)
Time Frame: Year 3
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Lap-Band
Number analyzed (Participants) | 87
kg/m^2 | 36 (8.94)

9. Secondary Outcome: Body Mass Index (BMI)
Time Frame: Year 4
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Lap-Band
Number analyzed (Participants) | 81
kg/m^2 | 36.39 (8.9)

10. Secondary Outcome: Body Mass Index (BMI)
Time Frame: Year 5
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Lap-Band
Number analyzed (Participants) | 74
kg/m^2 | 36.75 (8.98)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Lap-Band
All-Cause Mortality (participants affected / at risk) | 0/119
Serious Adverse Events (participants affected / at risk) | 24/119
Other Adverse Events (participants affected / at risk) | 99/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lap-Band (N=119)
Abdominal pannus (excess skin) (Gastrointestinal disorders) | 1
Band erosion (Gastrointestinal disorders) | 1
Band slippage (Gastrointestinal disorders) | 12
Cholecystitis (Gastrointestinal disorders) | 1
Cholelithiasis (Gastrointestinal disorders) | 2
Cholelithiasis (Aggravated) (Gastrointestinal disorders) | 1
Esophageal and gastric pouch dilatation (Gastrointestinal disorders) | 1
Gastric pouch dilatation (Gastrointestinal disorders) | 1
Left tibia surgery for Blount's disease (Musculoskeletal and connective tissue disorders) | 1
Nausea (General disorders) | 1
Perforated appendicitis (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Port leak (General disorders) | 2
Pregnancy with abortion (Pregnancy, puerperium and perinatal conditions) | 2
Right tibia surgery for Blount's disease (Musculoskeletal and connective tissue disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lap-Band (N=119)
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal subcutaneous infection (Gastrointestinal disorders) | 1
Abnormal EKG (junctional bradycardia) (Gastrointestinal disorders) | 1
Acne (Endocrine disorders) | 2
Acute dysphagia (General disorders) | 2
ADD (General disorders) | 2
ADHD (General disorders) | 1
Adnexal mass (Reproductive system and breast disorders) | 1
Adrenal Hyperplasia (General disorders) | 1
Anemia (General disorders) | 2
Anorexia (General disorders) | 1
Anxiety (Nervous system disorders) | 5
Anxiety Attack (Nervous system disorders) | 1
ARD (Acute Respiratory Failure) (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (General disorders) | 1
Band erosion (Gastrointestinal disorders) | 1
Band intolerance (Gastrointestinal disorders) | 2
Band intolerance (Chronic dysphagia) (Gastrointestinal disorders) | 1
Band slippage (Gastrointestinal disorders) | 9
Behavioural issue (General disorders) | 1
Bell's palsy (Musculoskeletal and connective tissue disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Chest pain (General disorders) | 1
Cholelithiasis (Gastrointestinal disorders) | 2
Chronic band intolerance (Gastrointestinal disorders) | 3
Chronic dysphagia with band tightening (Gastrointestinal disorders) | 1
Common cold (General disorders) | 6
Depression (General disorders) | 1
Depression (Aggravated) (General disorders) | 1
Device malfunction (Band aneurysm) (Gastrointestinal disorders) | 1
Dilated esophagus and gastric pouch (Gastrointestinal disorders) | 1
Dsyphagia (Musculoskeletal and connective tissue disorders) | 1
Dyslipidemia (Blood and lymphatic system disorders) | 1
Dyslipidemia (Aggravated) (Blood and lymphatic system disorders) | 3
Dysmenorrhea (Reproductive system and breast disorders) | 2
Dysphagia (General disorders) | 3
Dysphagia (ER visit) (General disorders) | 1
Ear and throat infection (Ear and labyrinth disorders) | 1
Eating disorder (Psychiatric disorders) | 1
Ecchymosis (post-op site) (Blood and lymphatic system disorders) | 1
Elevated bilirubin level (Blood and lymphatic system disorders) | 1
Elevated TSH (Respiratory, thoracic and mediastinal disorders) | 1
Elevated WBC (Blood and lymphatic system disorders) | 1
Endometriosis (General disorders) | 1
Epigastric pain (General disorders) | 1
Erosion on antrum (endoscopy) (Gastrointestinal disorders) | 1
Esophageal dilatation (General disorders) | 23
Esophageal irritation (General disorders) | 1
Esophageal pain (General disorders) | 1
Esophagitis (General disorders) | 6
Exacerbation of Eczema (Skin and subcutaneous tissue disorders) | 1
Excess skin (Skin and subcutaneous tissue disorders) | 2
Excess skin irritation (Skin and subcutaneous tissue disorders) | 1
Facial skin infection (Skin and subcutaneous tissue disorders) | 1
Fainting (General disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Flipped port (General disorders) | 1
Frozen pelvis (Renal and urinary disorders) | 1
Fungal infection (General disorders) | 1
Gallstones (General disorders) | 1
Gas pain (Gastrointestinal disorders) | 1
Gastric pouch dilatation (Gastrointestinal disorders) | 16
Gastric pouch dilation (Gastrointestinal disorders) | 5
Gastric pouch formation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastroenteritis (Gastrointestinal disorders) | 2
GE Reflux (General disorders) | 2
GERD (General disorders) | 2
Hair Thinning (General disorders) | 29
Headaches (General disorders) | 1
Heartburn (Gastrointestinal disorders) | 17
Hiatal hernia (Gastrointestinal disorders) | 1
Hiatal hernia (Esophagram) (Gastrointestinal disorders) | 1
HTN (Aggravated) (General disorders) | 1
Hyperbilirubinemia (General disorders) | 2
Hyperbilirubinemia (Aggravated) (General disorders) | 2
Hypercholesterolemia (Congenital, familial and genetic disorders) | 7
Hypercholesterolemia (aggravated) (Congenital, familial and genetic disorders) | 2
Hypertriglyceridemia (General disorders) | 1
Hypokalemia (General disorders) | 1
Hypothyroidism (General disorders) | 1
Influenza (Respiratory, thoracic and mediastinal disorders) | 1
Insomnia (Nervous system disorders) | 1
Iron deficiency (General disorders) | 2
Kidney stones (Gastrointestinal disorders) | 1
Knee injury (Left) (Musculoskeletal and connective tissue disorders) | 1
Leg cramps (Musculoskeletal and connective tissue disorders) | 1
Low Folate level (Blood and lymphatic system disorders) | 2
Low Hb level (Blood and lymphatic system disorders) | 3
Low iron level (General disorders) | 31
Low iron level (Aggravated) (General disorders) | 2
Low Vit. B12 level (General disorders) | 1
Low Vit. D level (General disorders) | 40
Low Vit. D level (Aggravated) (General disorders) | 12
Low Vit. D level (Baseline:24) (General disorders) | 1
Major depression (Cardiac disorders) | 1
Meniscus dislocation (Left) (Musculoskeletal and connective tissue disorders) | 1
Meniscus tear (Musculoskeletal and connective tissue disorders) | 1
Migraine (General disorders) | 3
Monocleosis (Immune system disorders) | 2
Mononucleosis (Immune system disorders) | 1
Multiple sclerosis (Nervous system disorders) | 1
Mumps (Infections and infestations) | 1
Narcotic addition (General disorders) | 1
Nausea (General disorders) | 1
Neck pain (General disorders) | 1
Numbness after exposing bright light (Immune system disorders) | 1
Panic attack (Nervous system disorders) | 1
Panic disorder (Nervous system disorders) | 1
Port leak (General disorders) | 1
Port protrusion (General disorders) | 1
Port site pain (General disorders) | 2
Post op site infection (General disorders) | 2
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Pregnancy with abortion (Pregnancy, puerperium and perinatal conditions) | 1
Proteinuria (Renal and urinary disorders) | 1
Psoriasis (Aggravated) (Immune system disorders) | 1
Reflux (Gastrointestinal disorders) | 17
Seasonal allergies (Immune system disorders) | 1
Self-inflicted forearm laceration (General disorders) | 1
Shoulder pain (General disorders) | 1
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 7
Stomach cramps (Gastrointestinal disorders) | 1
Strep throat (Respiratory, thoracic and mediastinal disorders) | 1
Suicidal threats (Psychiatric disorders) | 1
Testicular torsion (General disorders) | 1
Thrombocytopenia (Immune system disorders) | 2
Tooth pain (Immune system disorders) | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
Urinary tract infection (Renal and urinary disorders) | 4
Thrombocytopenia (small fat) (Blood and lymphatic system disorders) | 1
Viral gastroenteritis (Gastrointestinal disorders) | 2
Vit. D Deficiency (General disorders) | 5
Wound dehiscence (General disorders) | 1
Yeast infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT00587301/Prot_SAP_000.pdf